CLINICAL TRIAL: NCT06797635
Title: An Open-label Randomized Phase 2 Study to Evaluate Safety and Efficacy of Patritumab Deruxtecan Plus Pembrolizumab Administered Either Before or After Carboplatin/Paclitaxel Plus Pembrolizumab Compared With Pembrolizumab in Combination With Chemotherapy Followed by Surgery and Adjuvant Pembrolizumab for High-Risk Early-Stage Triple-Negative or Hormone Receptor-Low Positive/Human Epidermal Growth Factor Receptor-2 Negative Breast Cancer (HERTHENA-Breast03)
Brief Title: Study of Patritumab Deruxtecan Plus Pembrolizumab With Other Anticancer Agents in Participants With High-Risk Early-Stage Triple-Negative or Hormone Receptor-Low Positive/HER-2 Negative Breast Cancer (MK-1022-010, HERTHENA-Breast-03)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1022-010; MK-1022-010 (Other: MSD); 2024-514376-40-00 (Registry Identifier: EU CT); U1111-1307-7867 (Registry Identifier: UTN)
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan; pembrolizumab; Paclitaxel; Carboplatin; Doxorubicin; Epirubicin; Cyclophosphamide; Capecitabine; olaparib

STUDY DESIGN:
Intervention Model Description: Part 1 is non-randomized. Part 2 is randomized 1:1:1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin (Experimental): In Part 1, participants receive neoadjuvant pembrolizumab 200 mg via intravenous (IV) infusion every 3 weeks (Q3W) plus patritumab deruxtecan via IV infusion Q3W for 12 weeks, followed by pembrolizumab 200 mg via IV infusion Q3W plus paclitaxel 80 mg/m^2 via IV infusion every week (QW) and carboplatin AUC1.5 mg/ml/min via IV infusion QW for 12 weeks. At 3 to 6 weeks after last dose of neoadjuvant treatment, participants will undergo surgery for their breast cancer.
  Interventions: Biological: Patritumab deruxtecan; Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin
- Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin (Experimental): In Part 2, participants receive neoadjuvant pembrolizumab 200 mg IV infusion every Q3W plus patritumab deruxtecan (dose to be determined in part 1) IV infusion Q3W for 12 weeks, followed by pembrolizumab 200 mg IV infusion Q3W plus paclitaxel 80 mg/m^2 IV infusion QW and carboplatin AUC1.5 mg/ml/min IV infusion QW for 12 weeks. At 3-6 weeks after last dose of neoadjuvant treatment, participants undergo surgery for breast cancer. After surgery, participants receive adjuvant pembrolizumab 400 mg IV every 6 weeks (Q6W) for ~30 weeks. Additional adjuvant treatment of physician's choice (TPC) may be given to participants with residual disease. TPC options are olaparib 300 mg oral twice daily (BID) for 1 year (participants with germline BRCA mutation [gBRCAm] only), capecitabine 1000-1250 mg/m^2 oral BID days 1-14 and 22-35 Q6W for 4 six-week cycles or doxorubicin 60mg/m^2 (or epirubicin 90 mg/m^2) IV Q3W or every 2 weeks (Q2W) and cyclophosphamide 600 mg/m^2 IV Q3W or Q2W for 4 doses.
  Interventions: Biological: Patritumab deruxtecan; Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin hydrochloride; Drug: Epirubicin hydrochloride; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib
- Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan (Experimental): In Part 2, participants receive neoadjuvant pembrolizumab 200 mg IV infusion Q3W plus paclitaxel 80 mg/m^2 IV infusion QW and carboplatin AUC1.5 mg/ml/min IV infusion QW for 12 weeks, followed by pembrolizumab 200 mg IV infusion Q3W plus patritumab deruxtecan (dose to be determined in part 1) via IV infusion Q3W for 12 weeks. At 3 to 6 weeks after last dose of neoadjuvant treatment, participants will undergo surgery for their breast cancer. After surgery, participants will receive adjuvant pembrolizumab 400 mg IV infusion Q6W for ~30 weeks. Additional adjuvant TPC may be administered to participants with residual disease. TPC options include olaparib 300 mg oral BID for 1 year (participants with gBRCAm only), capecitabine 1000-1250 mg/m^2 oral BID days 1-14 and 22-35 Q6W for 4 six-week cycles or doxorubicin 60mg/m^2 (or epirubicin 90 mg/m^2) IV infusion Q3W or Q2W and cyclophosphamide 600 mg/m^2 IV infusion Q3W or Q2W for 4 doses.
  Interventions: Biological: Patritumab deruxtecan; Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin hydrochloride; Drug: Epirubicin hydrochloride; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib
- Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide (Active Comparator): In Part 2, participants receive neoadjuvant pembrolizumab 200 mg IV infusion Q3W plus paclitaxel 80 mg/m^2 IV infusion QW and carboplatin AUC1.5 mg/ml/min via IV infusion QW for 12 weeks, followed by pembrolizumab 200 mg IV infusion Q3W plus doxorubicin 60mg/m^2 (or epirubicin 90 mg/m^2) IV infusion Q3W and cyclophosphamide 600 mg/m^2 IV infusion Q3W for 12 weeks. At 3 to 6 weeks after last dose of neoadjuvant treatment, participants will undergo surgery for their breast cancer. After surgery, participants will receive adjuvant pembrolizumab 400 mg IV infusion Q6W for approximately 30 weeks. Additional adjuvant TPC may be administered to participants with residual disease. TPC options include olaparib 300 mg oral BID for 1 year (participants with gBRCAm only) or capecitabine 1000-1250 mg/m^2 oral BID days 1-14 and 22-35 Q6W for 4 six-week cycles.
  Interventions: Biological: Pembrolizumab; Drug: Paclitaxel; Drug: Carboplatin; Drug: Doxorubicin hydrochloride; Drug: Epirubicin hydrochloride; Drug: Cyclophosphamide; Drug: Capecitabine; Drug: Olaparib

INTERVENTIONS:
Biological: Patritumab deruxtecan — Administered via IV infusion as neoadjuvant treatment
  Other Names: MK-1022; HER3-DXd; U3-1402
  Arms: Part 1, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan
Biological: Pembrolizumab — Administered via IV infusion as neoadjuvant treatment in Part 1 and via IV infusion as neoadjuvant and adjuvant treatment in Part 2
  Other Names: MK-3475; KEYTRUDA®
Drug: Paclitaxel — Administered via IV infusion as neoadjuvant treatment
  Other Names: TAXOL®; ONXAL®
Drug: Carboplatin — Administered via IV infusion as neoadjuvant treatment
  Other Names: PARAPLATIN®
Drug: Doxorubicin hydrochloride — Administered via IV infusion as neoadjuvant treatment in Arm C and an option for adjuvant treatment for participants with residual disease in Arms A and B in Part 2
  Other Names: ADRIAMYCIN®
  Arms: Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan; Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide
Drug: Epirubicin hydrochloride — Administered via IV infusion as neoadjuvant treatment in Arm C and an option for adjuvant treatment for participants with residual disease in Arms A and B in Part 2
  Other Names: ELLENCE®
  Arms: Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan; Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide
Drug: Cyclophosphamide — Administered via IV infusion as neoadjuvant treatment in Arm C and an option for adjuvant treatment for participants with residual disease in Arms A and B in Part 2
  Other Names: CYTOXAN®
  Arms: Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan; Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide
Drug: Capecitabine — Administered via oral tablets as an option for adjuvant treatment for participants with residual disease in Part 2
  Other Names: XELODA®
  Arms: Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan; Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide
Drug: Olaparib — Administered via oral tablets as an option for adjuvant treatment for participants with germline BRCA mutations and residual disease in Part 2
  Other Names: LYNPARZA®
  Arms: Part 2, A: Pembrolizimab + patritumab deruxtecan → Pembrolizumab + paclitaxel + carboplatin; Part 2, B: Pembrolizumab + paclitaxel + carboplatin → Pembrolizumab + patritumab deruxtecan; Part 2, C: Pembro + paclitaxel + carboplatin→ Pembro + doxorubicin (or epirubicin) +cyclophosphamide

SUMMARY:
Researchers are looking for new ways to treat triple-negative breast cancer (TNBC) and hormone receptor (HR) low positive/human epidermal growth factor receptor-2 (HER2) negative breast cancer. The main goals of this study are to learn:

* About the safety of the study treatments and if people tolerate them
* If people who receive patritumab deruxtecan, pembrolizumab, and chemotherapy before surgery have fewer cancer cells removed during surgery compared to those who receive only pembrolizumab (pembro) and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has locally advanced, non-metastatic (M0), breast cancer, defined as any of the following combined primary tumor (T) and regional lymph node (N) staging per current American Joint Committee on Cancer (AJCC) criteria: cT1c, N1-N2; cT2, N0-N2; cT3, N0-N2; or cT4a-d, N0-N2
* Has centrally confirmed diagnosis of breast cancer that is triple-negative or HR-low+/HER2- breast cancer that will be treated according to the triple-negative breast cancer (TNBC) paradigm
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load
* Participants with a history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 28 days prior to allocation/randomization
* Has left ventricular ejection fraction (LVEF) of ≥50% or ≥ lower limit of normal (LLN) as assessed by echocardiogram (ECHO) or multigate acquisition scan (MUGA) scan

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has uncontrolled or significant cardiovascular disease before randomization
* Has clinically significant corneal disease
* Has human immunodeficiency virus (HIV) infection with a history of Kaposi sarcoma and/or multicentric Castleman disease
* Has received prior therapy with an anti-programmed death (PD)-1, anti-PD-L1, or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received any prior treatment, including radiation, systemic therapy, and/or definitive surgery for currently diagnosed breast cancer
* Has received prior treatment with an anti-human epidermal growth factor receptor 3 (HER3) antibody and/or antibody-drug conjugate (ADC) that consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g., trastuzumab deruxtecan)
* Has metastatic (Stage IV) breast cancer or cN3 nodal involvement
* Has known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease, or where suspected ILD/pneumonitis cannot be ruled out by standard diagnostic assessments
* Has an active infection requiring systemic therapy
* Has concurrent active HBV and HCV infection
* Has clinically severe respiratory compromise resulting from intercurrent pulmonary illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants Experiencing an Adverse Event (AE) | Up to ~43 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be presented for Part 1.
Part 1: Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLTs) | Up to 21 days
  A DLT is defined by the National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) Version 5.0, assessed by investigator as drug-related: Grade (gr) 3 or 4 nonhematologic toxicity (with exceptions); gr 3 or gr 4 laboratory values (with exceptions); gr 3 or 4 febrile neutropenia; prolonged delay (>2 weeks) in initiating Cycle 2 (cycle length = 3 weeks) due to intervention-related toxicity; any intervention-related toxicity that causes the participant to discontinue intervention during Cycle 1; interstitial lung disease as per investigator; any other gr ≥3 pulmonary toxicity; or gr 5 toxicity.
Part 1: Number of Participants who Discontinued Study Treatment Due to an AE | Up to ~30 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinued study treatment due to an AE will be presented for Part 1.
Part 2: Pathological Complete Response (pCR) Rate Using the Definition of ypT0/Tis ypN0 | Up to ~30 weeks
  pCR (ypT0/Tis ypN0) is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy at the time of definitive surgery.
Part 2: Number of Participants Experiencing an AE | Up to ~103 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who experience an AE will be presented for Part 2.
Part 2: Number of Participants who Discontinued Study Treatment Due to an AE | Up to ~90 weeks
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment. The number of participants who discontinued study treatment due to an AE will be presented for Part 2.

SECONDARY OUTCOMES:
Part 2: pCR-No Ductal Carcinoma in Situ (DCIS) Rate Using the Definition of ypT0 ypN0 | Up to ~30 weeks
  pCR-no DCIS (ypT0 ypN0) is defined as the absence of residual invasive and in situ cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes after completion of neoadjuvant systemic therapy at the time of definitive surgery.
Part 2: Event-Free Survival (EFS) | Up to ~100 months
  EFS is defined as the time from randomization to disease progression that precludes surgery, local or distant recurrence, or death due to any cause, whichever occurs first.
Part 2: Overall Survival (OS) | Up to ~100 months
  OS is defined as the time from randomization to date of death due to any cause.
Part 2: Distant Progression or Distant Recurrence-Free Survival (DPDRFS) | Up to ~100 months
  DPDRFS is defined as the time from randomization to first distant progression or distant recurrence event as assessed or death due to any cause, whichever occurs first.
Part 2: Residual Cancer Burden (RCB) | Up to ~30 weeks
  RCB is defined as residual disease in either the breast or lymph node at the time of surgery. RCB score provides a continuous measurement of the extent of residual cancer. There are four RCB classes: RCB-0 (RCB score 0), RCB-1 (0< RCB score <1.36), RCB-2 (1.36 <RCB score <3.28), and RCB-3 (RCB score >3.28).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (17):
- United States (8):
  - UCLA Hematology/Oncology - Parkside ( Site 0021), Santa Monica, California
  - Orchard Healthcare Research Inc. ( Site 0006), Skokie, Illinois
  - Intermountain Health St. Vincent Regional Hospital - Cancer Centers of Montana ( Site 0003), Billings, Montana
  - Northwest Cancer Specialists (Compass Oncology) ( Site 8003), Tigard, Oregon
  - SCRI Oncology Partners ( Site 7000), Nashville, Tennessee
  - Texas Oncology - DFW ( Site 8000), Dallas, Texas
  - Houston Methodist Hospital ( Site 0022), Houston, Texas
  - Virginia Oncology Associates (VOA) ( Site 8001), Norfolk, Virginia
- South Korea (3):
  - Seoul National University Hospital ( Site 2400), Seoul
  - Severance Hospital, Yonsei University Health System ( Site 2402), Seoul
  - Asan Medical Center ( Site 2401), Seoul
- Spain (3):
  - Institut Català d'Oncologia (ICO) - Badalona ( Site 1700), Badalona, Catalonia
  - Clinica Universidad de Navarra ( Site 1703), Madrid, Madrid, Comunidad de
  - Hospital Universitario Reina Sofia ( Site 1702), Córdoba
- Taiwan (3):
  - Taichung Veterans General Hospital ( Site 2502), Taichung
  - National Cheng Kung University Hospital ( Site 2503), Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 2501), Taipei

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com